CLINICAL TRIAL: NCT06157450
Title: A Phase I Single Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate Pharmacokinetics, Safety and Tolerability of ZSP1273 in Elder Participants
Brief Title: Pharmacokinetics of ZSP1273 in Elder Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ZSP1273-23-15
Record Dates: First submitted 2023-11-20; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Elder
MeSH Terms: interventions — ZSP1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: young participates (Experimental): 16 young participants(between 18~45 years old) will be given 600mg of ZSP1273.
  Interventions: Drug: ZSP1273
- Experimental:elder participates (Experimental): 16 elder participants(Age≥65 years old) will be given 600mg of ZSP1273.
  Interventions: Drug: ZSP1273

INTERVENTIONS:
Drug: ZSP1273 — Participants receive ZSP1273 orally.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and PK of ZSP1273 in elder Participants

ELIGIBILITY:
Inclusion Criteria:

1. Signature of a dated Informed Consent Form (ICF) indicating that the participates has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment.
2. Participants must be willing and able to adhere to the visit schedule and protocol requirements and be available to complete the study.
3. Body weight is no less than 50 kg in males and no less than 45 kg in females. Body mass index (BMI) 18≤BMI<28 kg/m2,BMI is determined by the following equation: BMI = weight/height2 (kg/m2).
4. Heart rate between 50-100 beats/min, Body temperature between 35.7-37.5℃

   Young Participants Only:
5. Participants must be ≥18 to ≤45 years old

   Elder Participants Only:
6. Participants must be ≥65 years old

Exclusion Criteria:

1. Participants with an allergic disposition (multiple drug and food allergies)
2. Participants who donated blood or bleeding profusely (> 400 mL) in the 3 months.
3. Participants with clinically significant disease, such as gastrointestinal disease, infection (e.g., respiratory or central nervous system infection), within 2 weeks before screening;
4. Participants who could not tolerate blood collection by venipuncture and/or had a history of dizzy with blood and needles

   Young Participants Only:
5. Participants had taken or planned to take any prescription medication, over-the-counter medication, vitamin product, or herbal medicine within 2 weeks before screening;
6. Physical examination, vital signs, laboratory tests (blood routine +CRP, urine routine + urine sediment, blood biochemistry, coagulation function, infectious disease test, glycosylated hemoglobin test), 12-lead electrocardiogram, chest CT, abdominal color Doppler ultrasound and other examinations have clinical significance

   Elder Participants Only:
7. Participants had a history of or evidence of cardiovascular disease before screening: uncontrolled hypertension, orthostatic hypotension, severe arrhythmia, heart failure, Adams-stokes syndrome, unstable angina, myocardial infarction within the past 6 months before screening, or history of tachycardia/bradycardia requiring medical treatment, and degree II-III atrioventricular block.
8. Participants who had other serious organ-systemic serious diseases at screening, including but not limited to respiratory, neurologic, hematologic, endocrine, oncologic, immunologic, psychiatric, or cardio-cerebrovascular diseases, and was judged by the investigator to be ineligible for participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 to Day 5
  The Cmax of a single dose of ZSP1273 in elder participants and young participates will be evaluated and compared.
Area under the concentration-time curve from time zero to infinity (AUCinf) | Day 1 to Day 5
  The AUCinf of a single dose of ZSP1273 in elder participants and young participates will be evaluated and compared.
Area under the concentration-time curve from time zero to last time of quantifiable concentration (AUClast) | Day 1 to Day 5
  The AUClast of a single dose of ZSP1273 in elder participants and young participates will be evaluated and compared.

SECONDARY OUTCOMES:
Number of participants with drug-related adverse events as assessed by CTCAE v5.0 | Day 1 to Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided